CLINICAL TRIAL: NCT00360750
Title: A Data Collection Study to Compare the Outcome for Children With Advanced Unilateral Retinoblastoma Treated With or Without Post-Enucleation Chemotherapy ± Radiotherapy on RB 2005 11 With Historical Controls Receiving no Additional Therapy
Brief Title: Chemotherapy With or Without Radiation Therapy or Observation in Treating Young Patients With Advanced Retinoblastoma Who Have Undergone Surgery to Remove the Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000481598; CCLG-RB-2005-11; EU-20616; EUDRACT-2004-001367-21
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Retinoblastoma
Keywords: intraocular retinoblastoma; extraocular retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Carboplatin; Cytarabine; Etoposide; Vincristine; Watchful Waiting; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cytarabine
Drug: etoposide
Drug: vincristine sulfate
Other: clinical observation
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, vincristine, etoposide, and cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy with or without radiation therapy after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor does not need more treatment until it progresses. In this case, observation may be sufficient.

PURPOSE: This clinical trial is studying how well chemotherapy with or without radiation therapy or observation works in treating young patients with advanced retinoblastoma who have undergone surgery to remove the eye.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare outcome data in children with advanced unilateral retinoblastoma with historical controls in order to determine whether post-enucleation chemotherapy with or without radiotherapy improves outcome.
* Determine the disease-free and overall survival of children with unilateral retinoblastoma with no adverse histological features who undergo observation after enucleation.
* Determine the toxicity of these regimens in these patients.

OUTLINE: This is a nonrandomized study. Patients are assigned to 1 of 3 treatment groups according to histological features.

* Group 1 (no adverse histological features): Patients are observed and monitored for the development of orbital recurrence and metastatic disease.
* Group 2a (deep choroidal invasion and/or retrolaminar invasion of the optic nerve and disease in the anterior chamber): Patients receive carboplatin IV over 1 hour, vincristine IV, and etoposide IV over 4 hours on day 1, and, if necessary, intrathecal cytarabine on day 2. Treatment repeats every 21 days for 4 courses.
* Group 2b (invasion of the cut end of the optic nerve): Patients receive carboplatin IV over 1 hour, vincristine IV, and etoposide IV over 4 hours on day 1, and, if necessary, intrathecal cytarabine on day 2. Treatment repeats every 21 days for 6 courses. Patients also undergo orbital radiotherapy 5 days a week for 4 weeks.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unilateral retinoblastoma

  * Prior primary enucleation required
* No metastatic spread

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy
* No concurrent steroids as antiemetic agents

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-09; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Outcome data compared to historical controls
Disease-free and overall survival in children undergoing observation after enucleation
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Helen Jenkinson, MD, Study Chair — Birmingham Children's Hospital
Locations (13):
- United Kingdom (13):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Queen's Medical Centre, Nottingham, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland